CLINICAL TRIAL: NCT00044967
Title: A Prospective Study Of The Prognostic Significance Of Microsatellite Instability In Patients With Early Age-Of-Onset Colorectal Cancer
Brief Title: Genetic Study of Young Patients With Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACOSOG-Z0190; ACOSOG-Z0190; CDR0000069465 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients undergo baseline colonoscopy before or within 6 months of initial curative resection and then surveillance colonoscopy at 1, 3, and 5 years (+/- 6 months) after resection. The number, size, location, histology, and method of removal of polyps are documented at the time of colonoscopy. Patients also undergo microsatellite instability (MSI) status testing and complete family history questionnaires at baseline.
  The prognostic significance of family history and MSI status is evaluated. The individual histologic features of the tumors are compared with the MSI status to determine their predictive value. The histologic features are also correlated with outcome to determine their prognostic significance.
  Patients may be referred for genetic counseling.
  Interventions: Genetic: microsatellite instability analysis

INTERVENTIONS:
Genetic: microsatellite instability analysis

SUMMARY:
RATIONALE: Identifying gene mutations (microsatellite instability) may allow doctors to plan effective treatment for patients who develop colorectal cancer at an early age.

PURPOSE: Genetic trial to determine the significance of gene mutations in helping predict the outcome of treatment in patients who develop stage I, stage II, or stage III colorectal cancer at an early age.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the prognostic significance (e.g., overall survival) of microsatellite instability (MSI) status in patients with early age-of-onset stage I-III colorectal cancer, assuming the presence of a quantitative interaction between MSI status and family history of cancer.
* Evaluate the development of metachronous neoplasms in this patient population.
* Evaluate the histologic features and genetic changes associated with hereditary nonpolyposis colorectal cancer in this patient population.

OUTLINE: This is a multicenter study. Patients are stratified according to family history using the Amsterdam II criteria for hereditary nonpolyposis colorectal cancer (positive vs negative).

Patients undergo baseline colonoscopy before or within 6 months of initial curative resection and then surveillance colonoscopy at 1, 3, and 5 years (+/- 6 months) after resection. The number, size, location, histology, and method of removal of polyps are documented at the time of colonoscopy. Patients also undergo microsatellite instability (MSI) status testing and complete family history questionnaires at baseline.

The prognostic significance of family history and MSI status is evaluated. The individual histologic features of the tumors are compared with the MSI status to determine their predictive value. The histologic features are also correlated with outcome to determine their prognostic significance.

Patients may be referred for genetic counseling.

A certificate of confidentiality protecting the identity of research participants in this project has been issued by the National Cancer Institute.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage I-III adenocarcinoma of the colon or rectum
* Must have undergone an initial curative resection within the past year

  * No colon or rectal cancer resection that does not allow for definitive T or N staging
  * No initial post-surgical surveillance colonoscopy prior to study entry
* Must have a pathology specimen, with representative normal and tumor tissues, available for submission to the ACOSOG Central Specimen Bank prior to study entry
* No personal or family history of familial adenomatous polyposis
* No recurrent colorectal cancer

PATIENT CHARACTERISTICS:

Age

* 18 to 49 at first diagnosis

Other

* Must be willing to provide a family cancer history to the study team and continue with follow-up colonoscopic surveillance
* No other malignancy within the past 5 years except completely resected cervical cancer or nonmelanoma skin cancer
* No evidence of recurrence of other prior malignancy

PRIOR CONCURRENT THERAPY:

Radiotherapy

* No prior pelvic radiotherapy for rectal cancer
* No concurrent preoperative pelvic radiotherapy for rectal cancer

Surgery

* See Disease Characteristics

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with adenocarcinoma of the colon or rectum.
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2002-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose G. Guillem, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (73):
- United States (71):
  - Providence Cancer Center, Mobile, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arrowhead Regional Medical Center, Colton, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Morton Plant Hospital, Clearwater, Florida
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Surgical Oncology of Northeast Georgia, Gainesville, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush Copley Medical Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Great Lakes Cancer Institute - McLaren, Flint, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Digestive Health Specialists, P.A., Tupelo, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Cancer Center at Creighton University Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Akron General's McDowell Cancer Center, Akron, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Integris Oncology Services, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Sarah Cannon Cancer Center at Parkridge Medical Center, Chattanooga, Tennessee
  - Baptist Cancer Institute at Baptist Memorial Hospital - Memphis, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Baptist Hospital, Nashville, Tennessee
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - INOVA Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Associated Surgeons P.S., Spokane, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Fox Valley Surgical Associates at Appleton Medical Center, Appleton, Wisconsin
  - Appleton Medical Center, Appleton, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (2):
  - Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario